CLINICAL TRIAL: NCT05188014
Title: Effects of the Menstrual Cycle on Blood Glucose Changes During Exercise in Women With Type 1 Diabetes Using Oral Contraceptives
Brief Title: Exercise and the Menstrual Cycle in Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro0083867
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will be in a single study arm.
  Interventions: Behavioral: Luteal Phase Aerobic Exercise; Behavioral: Follicular Phase Aerobic Exercise

INTERVENTIONS:
Behavioral: Luteal Phase Aerobic Exercise — Participants will perform 45 minutes of moderate (60% VO2peak) aerobic exercise on a cycle ergometer during the last week of active pill consumption.
Behavioral: Follicular Phase Aerobic Exercise — Participants will perform 45 minutes of moderate (60% VO2peak) aerobic exercise on a cycle ergometer within 5 days of starting their menses.

SUMMARY:
Female participants with type 1 diabetes using oral contraceptives will be asked to wear a continuous glucose monitor for at least three days on two separate occasions (once during the last week of active pills and once during the no pill/placebo pill phase of the menstrual cycle). An exercise session (45 minutes of aerobic exercise at 60% VO2peak on a cycle ergometer) will take place at 5 pm on the second day of glucose monitoring.

DETAILED DESCRIPTION:
Pre-test measures: Interested participants will be invited to the Physical Activity and Diabetes Laboratory on the main campus of the University of Alberta. They will be asked questions related to their menstrual cycle, physical activity levels and medication. Blood pressure will also be measured to assess their eligibility. Where participants are eligible, anthropometric characteristics will be measured using standard protocols. A blood sample will be drawn for assessment of HbA1c. Participants will perform an incremental treadmill test to volitional exhaustion. Indirect calorimetry will be used to assess oxygen consumption and carbon dioxide production to determine the participant's aerobic capacity.

Testing sessions: Participants will perform two testing sessions separated by at least 5 days. One session will take place during the last week of active pill consumption of monophasic hormonal contraceptives. The second session will take place during the placebo pill consumption phase (i.e. menses). Participants will be asked to arrive at the lab at around 4:00 pm for both sessions, which will be randomly assigned. During the sessions, participants will be asked to perform 45 minutes of aerobic exercise on an ergonomic cycle ergometer at 60% of the participant's pre-determined aerobic capacity. Blood samples will be drawn at baseline, at the end of exercise, and an hour post-exercise via an IV catheter. Participants will be asked to match their daily food and insulin intake as closely as possible from one testing session to the next for the day before, day of and day after the testing session. They will also be asked to avoid strenuous exercise and alcohol intake.

A continuous glucose monitor (CGM) sensor will be subcutaneously inserted by one of the investigators (trained by a group from the CGM manufacturer) into the anterior abdominal area of the participant in the morning of the day prior to each testing session. The participant will wear the CGM for at least 24 hours before the exercise session, and at least 24 hours after the exercise session.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes diagnosed for at least 1 year
* regular menses
* using monophasic oral contraceptives
* residing in Edmonton, Alberta and able to visit the lab at the University of Alberta

Exclusion Criteria:

* HbA1c > 9.9%
* frequent and unpredictable hypoglycemia
* change in insulin management strategy within two months of the study
* use of an automated insulin delivery system
* blood pressure > 140/95
* history of cardiovascular disease
* severe peripheral neuropathy
* active proliferative retinopathy
* use of medications (other than insulin) that would affect blood glucose levels
* any musculoskeletal condition that would contraindicate exercise (e.g. sprain, strain, joint injury, etc.)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | Pre-exercise (0 minutes), post-exercise (45 minutes) and 1 hour post-exercise
  Change in blood glucose, with samples drawn via IV catheter

SECONDARY OUTCOMES:
Interstitial glucose (continuous glucose monitoring) | 6 hours, 12 hours, overnight (midnight to 6 am) and 24 hours post-exercise
  Mean CGM glucose
coefficient of variation (CV) | 6 hours, 12 hours, overnight (midnight to 6 am) and 24 hours post-exercise
  measure of variability for continuous glucose monitoring data
standard deviation (SD) | 6 hours, 12 hours, overnight (midnight to 6 am) and 24 hours post-exercise
  measure of variability for continuous glucose monitoring data
frequency of hypoglycemia | 6 hours, 12 hours, overnight (midnight to 6 am) and 24 hours post-exercise
  number of times that CGM glucose is equal to or lower than 3.9 mmol/L
frequency of hyperglycemia | 6 hours, 12 hours, overnight (midnight to 6 am) and 24 hours post-exercise
  number of times that CMG glucose is equal to or greater than 10.0 mmol/L
percent of time in range | 6 hours, 12 hours, overnight (midnight to 6 am) and 24 hours post-exercise
  percent of time with CGM glucose between 4.0 and 9.9 mmol/L
percent of time in hypoglycemia | 6 hours, 12 hours, overnight (midnight to 6 am) and 24 hours post-exercise
  amount of time spent with CGM glucose equal to or less than 3.9 mmol/L
percent of time in hyperglycemia | 6 hours, 12 hours, overnight (midnight to 6 am) and 24 hours post-exercise
  amount of time spent with CGM glucose equal to or greater than 10.0 mmol/L

OTHER OUTCOMES:
Carbohydrate supplementation | Between 0 minutes and 45 minutes (during exercise)
  Grams of carbohydrate provided to prevent hypoglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Diabetes Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No